CLINICAL TRIAL: NCT05645822
Title: Screen and Treat Implementation in Insecure Areas With Limited Capacities for HAT Control
Brief Title: Screen and Treat Implementation for HAT Control
Status: Withdrawn | Type: Observational
Why Stopped: There is a problem with the provision of the treatment, we are unable to provide sufficient number of treatments for the study participants
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); SANRU Asbl, Soins de Santé Primaires en Milieu Rural, République Démocratique du Congo (Unknown); Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: Screen&treat
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Sleeping Sickness; Trypanosomiasis, African
Keywords: Sleeping sickness; Human African Trypanosomiasis; Fexinidazole
MeSH Terms: conditions — Trypanosomiasis, African

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples from sero-positive study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with symptoms attributable to gHAT: The study will include any person that attends any of the participating healthcare facilities with symptoms that could be attributed to gHAT (long-term fever (unless other obvious causes), headache for a long period (more than 14 days), presence of enlarged lymph nodes in the neck, severe weight loss, weakness, pruritus, amenorrhea, abortions or sterility, psychiatric problems (aggressiveness, apathy, mental confusion, anxiety), sleep disturbances, motor weakness, logorrhea, speech impairment, ataxia, abnormal gait, abnormal movements or seizures) and accepts to participate.
  Interventions: Other: Screen&treat

INTERVENTIONS:
Other: Screen&treat — Study participants will be tested with an RDT to prove the presence of antibodies against Trypanosoma brucei gambiense. Should the RDT be positive, they will be offered the 10-day treatment with fexinidazole, and an additional blood sample will be taken for the post hoc confirmation of the disease.

SUMMARY:
Human African Trypanosomiasis (HAT), or sleeping sickness, is one of the parasitic diseases targeted for interruption of transmission by 2030 by the WHO. The development of fexinidazole as treatment is a huge step towards this achievement; however, the diagnostic algorithm remains complex due to limited sensitivity and specificity of the available tests. A combination of serological screening and confirmation of infection through parasite visualization remains the preferred strategy, although it can be difficult to ensure its full performance in areas that are hard to reach or have limited access to electricity and other means.

The present study would like to test an approach of ensuring treatment with fexinidazole of sero-suspects without confirmation of disease, among patients that consult fixed health infrastructures in the provinces of Maniema, Lomami and Tanganyika. This should enable access to gHAT treatment for patients living in hard to reach areas, actively seeking health care.

DETAILED DESCRIPTION:
In this study, all gHAT suspects that attend participating health facilities with suggestive symptoms and test positive in an antibody detection rapid test, will presumptively be treated with fexinidazole. Blood samples will be collected for the post-hoc confirmation of the infection. Nine Health facilities have been selected in the health zones of Kasongo, Kibombo, Kunda and Samba (province of Maniema), Kongolo (province of Tanganyika) and Lubao (province of Lomami) by the PNLTHA, and ITM, based on both epidemiological data and operational considerations.

All patients that consult the selected facilities showing any symptom that could be attributed to gHAT will be offered to participate in the study and kindly requested to provide informed consent. Participants will be tested using the rapid diagnostic test (RDT) HAT Sero-K-SeT. All positive individuals will be asked to provide a venous blood sample, that will be sent to the Institut National de Recherche Biomédical (INRB) or Centre de Recherche en Santé de Kimpese (CRSK) for further serological testing with iELISA and/or immune trypanolysis (TL) and to confirm diagnosis with molecular testing. They will also be offered a 10-day fexinidazole treatment, as inpatient. After treatment, the study participants will be asked to return to the health facility after six months for a clinical follow-up.

Two follow -up visits (3 and 6 months) will be actively organized for all patients with a positive result in iELISA and/or molecular tests conducted at INRB/Kimpese laboratory, through active tracing by health facilities and community members. At the 3 month visit, a clinical examination and DNA/RNA sampling for molecular testing will be performed. At the 6 month visit, adverse events and disease status will be assessed based on clinical signs or symptoms. After the 6-month visit, all patients with a confirmed gHAT infection will be invited to come back to health facility 12, 18 and 24 months after treatment, following WHO guidelines, to confirm cure.

ELIGIBILITY:
Inclusion Criteria:

* Show any suggestive symptoms of gHAT, such as headache (>14 days), long-term fever unless other obvious cause(s), malaise, weakness, arthralgia, facial edema, pruritus, lymphadenopathy, weight loss, mental confussion, abnormal behavior, logorrhea, speech impairment, anxiety, tremor, motor weakness, ataxia, abnormal gait, abnormal movements or seizures;
* Being older than 6 years old and weighing at least 20 kg;
* Willing and able to provide written informed consent (assent for minors);
* Minors (6 to 17 years old) willing and able to provide a written assent, after obtaining written informed consent from their parents.

Exclusion Criteria:

* Being younger than 6 years old or weighing less than 20 kg;
* Refusal to provide informed consent;
* Previously treated for HAT (questionnaire to patients and/or family members);
* Pregnant women.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 9 health facilities in the endemic health zones of Kasongo, Kikombo, Kunda and Samba in the province of Maniema, Kongolo in the province of Tanganyika and Lubao in the province of Lomami are selected based on reported HAT cases 3 years prior, where fexinidazole treatment has been provided through PNLTHA or DNDi and where sample transport will be ensured by the NGO SANRU, despite difficult accessibility.
  The study aims to include every person that attends the participating fixed healthcare facilitie with suggestive symptoms of gHAT (see above) and is willing to provide informed consent. Since the feasibility of this approach is being tested, as many participants as possible will be included from the pool of people that attend participating healthcare centers during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility of an alternative operational approach for the diagnosis and treatment of gHAT patients in areas with limited access and diagnostic capacities. | 11 months
  This qualitative study will assess:
  * Number of people with suggestive symptoms;
  * Number of participants that test positive in the rapid diagnostic test;
  * Number of sero-positive individuals who accept fexinidazole treatment and
  * Number of treated individuals who test positive in further serological/molecular tests.

SECONDARY OUTCOMES:
Assess gHAT transmission in the provinces of Maniema, Tanganyka and partially Lomami. | 11 months
  Based on the number of sero-positive individuals and confirmed infections, calculate gHAT incidence in the study areas.
Contribute to the collection of evidence of the use of fexinidazole. | 11 months.
  The frequency and severity of any adverse effect due to the fexinidazole treatment will be recorded by a healthcare professional during the 10-day regime as well as in the 6-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Inocencio da Luz, PhD, Principal Investigator — Institute of Tropical Medicine

IPD SHARING:
Plan to Share IPD: Undecided